CLINICAL TRIAL: NCT01579019
Title: A Study of RO5024048 in Combination With Ritonavir-Boosted Danoprevir and Pegasys/Copegus in Patients With Chronic Hepatitis C Genotype 1 Who Have Failed Prior HCV Protease Inhibitor Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV22877; 2010-022659-41 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir; peginterferon alfa-2a; Ribavirin; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1000 mg 24 weeks (Active Comparator)
  Interventions: Drug: RO5024048; Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]
- 1000 mg 26 weeks (Active Comparator)
  Interventions: Drug: RO5024048; Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]; Drug: ritonavir
- 1500 mg 24 weeks (Experimental)
  Interventions: Drug: RO5024048; Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]; Drug: ritonavir
- 1500 mg 26 weeks (Experimental)
  Interventions: Drug: RO5024048; Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]; Drug: ritonavir

INTERVENTIONS:
Drug: RO5024048 — 1500 mg po bid, 24 or 26 weeks
  Arms: 1500 mg 24 weeks; 1500 mg 26 weeks
Drug: RO5024048 — 1000 mg po bid, 24 or 26 weeks
  Arms: 1000 mg 24 weeks; 1000 mg 26 weeks
Drug: danoprevir — 100 mg po bid, Weeks 1 to 24 or Weeks 3 to 26
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc qw, 24 or 26 weeks
Drug: ribavirin [Copegus] — 1000 mg or 1200 mg po daily, 24 or 26 weeks
Drug: ritonavir — 100 mg po bid, Weeks 1 to 24 or Weeks 3 to 26
  Arms: 1000 mg 26 weeks; 1500 mg 24 weeks; 1500 mg 26 weeks

SUMMARY:
This randomized, double blind, phase II study will evaluate the efficacy and safety of two doses of RO5024048 in combination with ritonavir-boosted danoprevir and Pegasys (peginterferon alpha-2a) and Copegus (ribavirin) in patients who failed a prior protease inhibitor containing regimen with or without pegylated interferon. Patients will be randomized to receive either a 2-week lead-in of RO5024048 (1500 mg or 1000 mg orally twice daily) in combination with Pegasys (180 mcg subcutaneously weekly) and Copegus (1000 mg or 1200 mg orally daily) followed by 24 weeks of therapy with RO5024048 in combination with danoprevir (100 mg orally twice daily) plus ritonavir (100 mg orally twice daily) and Pegasys and Copegus (QUAD therapy), or 24 weeks of therapy with RO5024048 in combination with danoprevir plus ritonavir and Pegasys and Copegus (QUAD therapy). Anticipated time on study treatment is 24 or 26 weeks, with a treatment-free follow-up of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Hepatitis C genotype 1 infection
* Serum HCV quantifiable by Roche COBAS TaqMan HCV Test v2.0
* Liver biopsy (within 24 months) or Fibroscan (within 12 months) before first administration of study drug consistent with chronic hepatitis C and demonstrating absence of liver cirrhosis
* Documented failed prior treatment with protease inhibitor (evidenced by viral breakthrough or partial response while on treatment or relapse after treatment), including documentation on treatment with other direct-acting antiviral agents and other HCV antiviral treatment
* Patients must have discontinued prior HCV treatment at least 24 weeks prior to first dose of study drug in this trial

Exclusion Criteria:

* Infection with any HCV genotype other than genotype 1
* Evidence of any variants associated with protease inhibitor resistance at screening
* Body mass index (BMI) <18 or >/=36 kg/m2
* Positive for hepatitis A or hepatitis B infection
* Use of any systemic antiviral therapy with perceived activity against HCV </=1 month prior to first dose of study drug
* History or evidence of a medical condition associated with chronic liver disease other than chronic hepatitis C
* Pregnant or breastfeeding women
* Males with female partners who are pregnant
* History of immunologically mediated disease; patients with rheumatoid arthritis requiring only intermittent non-steroidal anti-inflammatory medications or with celiac disease will be allowed
* History or evidence of decompensated liver disease
* History or evidence of renal disease; patients with history of nephrolithiasis will be allowed
* Uncontrolled Type 1 or 2 diabetes
* History or evidence of chronic pulmonary disease associated with functional limitation
* History of severe cardiac disease History of any neoplastic disease within the last 5 years, except for localized or in situ carcinoma of the skin (e.g. basal or squamous cell carcinoma)
* Evidence of excessive alcohol, drug or substance abuse (excluding marijuana use) within 1 year of the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response (defined as unquantifiable serum HCV RNA) 12 weeks after treatment (SVR-12) | approximately 2 years

SECONDARY OUTCOMES:
Sustained virologic response 4 weeks after treatment (SVR-4) | approximately 2 years
Sustained virologic response 24 weeks after treatment (SVR-24) | approximately 2 years
Change in serum HCV RNA levels | from baseline to Week 12
Virologic response over time | from baseline to 24 weeks after treatment
Correlation between trough concentrations of RO4995855 and virologic response | approximately 2 years
Incidence of direct-acting antiviral (DAA) resistance, including re-emergence of protease inhibitor resistant virus | approximately 2 years
Safety: Incidence of adverse events | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche